CLINICAL TRIAL: NCT03478930
Title: Open-Label Extension Study of Omalizumab in Patients With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: An Extension Study of Omalizumab in Participants With Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA40169; 2017-003450-16 (EudraCT Number)
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Nasal Polyps; Chronic Rhinosinusitis
MeSH Terms: conditions — Nasal Polyps | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Although this is an open-label study and all participants will be receiving omalizumab, in order to minimize bias in this study participants and the evaluating physicians will be blinded to treatment assignment of the previous studies (GA39688/GA39855) until all participants have either completed the study through the follow-up period (Week 76) or discontinued early from the study, the database is locked, and the study analyses are final.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Study GA39688 Omalizumab (Experimental): Participants who received omalizumab once every 2 weeks (Q2W) or once every 4 weeks (Q4W) in Study GA39688 will continue to receive omalizumab at Week 24 at the same dosing schedule.
  Interventions: Drug: Omalizumab
- Cohort A: Study GA39688 Placebo (Experimental): Participants who received placebo Q2W or Q4W in Study GA39688 will start receiving omalizumab Q2W or Q4W at Week 24 at the same dosing schedule.
  Interventions: Drug: Omalizumab; Drug: Placebo
- Cohort B: Study GA39855 Omalizumab (Experimental): Participants who received omalizumab Q2W or Q4W in Study GA39855 will continue to receive omalizumab at Week 24 at the same dosing schedule.
  Interventions: Drug: Omalizumab
- Cohort B: Study GA39855 Placebo (Experimental): Participants who received placebo Q2W or Q4W in Study GA39855 will start receiving omalizumab Q2W or Q4W at Week 24 at the same dosing schedule.
  Interventions: Drug: Omalizumab; Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab will be administered as a subcutaneous (SC) injection Q2W or Q4W.
  Other Names: Xolair
Drug: Placebo — Participants will not be receiving placebo in this OLE study. Participants who were randomized to the placebo arms for 24 weeks in studies GA39688/GA39855 and then enter this OLE study will receive omalizumab, but they will be placed in separate analysis cohorts.
  Arms: Cohort A: Study GA39688 Placebo; Cohort B: Study GA39855 Placebo

SUMMARY:
The overall purpose of this study is to evaluate the safety, efficacy, and durability of response of omalizumab in an open-label setting in adult participants with chronic rhinosinusitis with nasal polyps who completed the double-blind, placebo-controlled, Phase III studies GA39688 (NCT03280550) or GA39855 (NCT03280537). Participants will be eligible for enrollment in the study at, or within 28 days after, the Week 24 visit of Studies GA39688/GA39855. After enrollment into this open-label extension (OLE) study, participants will receive 28 weeks of dosing of omalizumab before entering a 24-week off-treatment observation phase of the study. Baseline in this OLE study is defined as the last pre-treatment measurement prior to randomization in Studies GA39688/GA39855 (i.e., baseline of Studies GA39688/GA39855). The data that will be reported from baseline to Week 24 inclusive will come from Studies GA39688/GA39855.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Participation in Study GA39688 or GA39855, including completion of endoscopy and other assessments at Week 24, without discontinuation of study drug
* Completion of eDiary daily assessments for at least 4 out of 7 days in the week prior to the Week 24 visit of Study GA39688 or GA39855
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods during the treatment period and for 60 days after the last dose of study drug

Exclusion Criteria:

* Anaphylaxis/hypersensitivity related to study drug in Study GA39688 or GA39855
* Serious adverse events related to study drug in Study GA39688 or GA39855 that the investigator or Sponsor determines may jeopardize the patient's safety if he or she continues in the study
* Uncontrolled epistaxis within Study GA39688 or GA39855
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 60 days after the last dose of omalizumab
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (79):
- United States (25):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Jonathan Corren MD, Inc., Los Angeles, California
  - The Allergy Station at Sacramento ENT, Roseville, California
  - Bensch Clinical Research LLC, Stockton, California
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Specialist Global Research, Hialeah, Florida
  - Vitae Research Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Asthma & Allergy of Idaho, Twin Falls, Idaho
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Chesapeake Clinical Research Inc - CRN, Baltimore, Maryland
  - Institute for Asthma & Allergy, Chevy Chase, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Missouri Health Care System, Columbia, Missouri
  - Northwell Health, Great Neck, New York
  - Montefiore Medical Center, The Bronx, New York
  - Vital Prospects Clinical Research Institute PC - CRN, Tulsa, Oklahoma
  - Allergy Associates Research Center LLC - CRN, Portland, Oregon
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - TTS Research, Boerne, Texas
  - Allergy & Asthma Res Ctr PA, San Antonio, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (2):
  - Yang Medicine, Ottawa, Ontario
  - Hopital du Saint Sacrement, Québec, Quebec
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Chirurgicka klinika, Hradec Králové
  - Stredomoravska nemocnicni a.s. - odstepny zavod Nemocnice Prostejov, Prostějov
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux Hopital Pellegrin, Bordeaux
  - Hopital de Hautepierre, Strasbourg
  - Nouvel Hopital Civil; Pole de Pathologie Thoracique, Strasbourg
- Germany (3):
  - Charie Campus Mitte; Hals, Nasen, Ohrenheilkunde, Berlin
  - Universitatsklinikum Leipzig, Leipzig
  - Universitatsklinikum Schleswig-Holstein; Klinik fuer Innere Medizin I, Lübeck
- Hungary (4):
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Szent Imre Egyetemi Oktatokorhaz, Budapest
  - Szent Janos Korhaz es Eszak-Budai Egyesitett Korhazak, Budapest
  - Pecsi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Pécs
- Mexico (2):
  - Unidad de Investigacion CIMA SC, Chihuahua City
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
- Poland (12):
  - Synexus Affiliate - Clinic Med s.j. Bialystok, Bialystok
  - Synexus - Gdynia, Gdynia
  - Synexus - Katowice, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Medyczne ALL-MED, Krakow
  - Centrum Medyczne Wos i Piwowarczyk, Krakow
  - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin
  - Synexus - Poznan, Poznan
  - Synexus - Warsaw, Warsaw
  - Centrum Medyczne Biotamed, Wieliczka
  - Synexus - Wroclaw, Wroclaw
  - EMC Instytut Medyczny S.A., Wroclaw
- Portugal (4):
  - Centro Hospitalar do Baixo Vouga E.P.E. - Hospital de Aveiro; Servicos Farmaceuticos, Aveiro
  - Hospital de Braga, Braga
  - Hospital Senhora da Oliveira - Guimarães, E.P.E, Guimarães
  - Centro Hospitalar do Algarve - Hospital de Portimao, Portimão
- Russia (4):
  - Central Clinical Hospital With Polyclinic of President Administration of RF, Moscow, Moscow Oblast
  - Medical Center Uromed, Smolensk, Moscow Oblast
  - LLC Kurator, Saint Petersburg, Sankt-Peterburg
  - Terapharm, Llc, Stavropol
- Spain (6):
  - Hospital de Jerez, Jerez de la Frontera, Cadiz
  - CHUS - H. Clinico U. de Santiago; Servicio de Farmacia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (8):
  - Municipal Health Care Institution Regional clinical specialized dispensary of radiation protection, Kharkiv, Kharkiv Governorate
  - State Institution Institute of Otolaryngology n.a. Prof. O.S., Kyiv, KIEV Governorate
  - Ternopil Municipal City Hospital, Ternopil, Podolia Governorate
  - Municipal Institution "City Clinical Hospital #3", Zaporizhzhia, Polissya Okruha
  - University Clinic, Ivano-Frankivsk, Poltava Governorate
  - Poltava Regional Clinical Hospital n.a. M.V. Skliphosovskyi, Poltava, Poltava Governorate
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Kyiv City Clinical Hospital #9, Kyiv
- Wigan,Wrighington & Leigh NHS Trust, Wigan, United Kingdom

REFERENCES:
- [Derived] Gevaert P, Mullol J, Saenz R, Ko J, Steinke JW, Millette LA, Meltzer EO. Omalizumab improves sinonasal outcomes in patients with chronic rhinosinusitis with nasal polyps regardless of allergic status. Ann Allergy Asthma Immunol. 2024 Mar;132(3):355-362.e1. doi: 10.1016/j.anai.2023.11.001. Epub 2023 Nov 10. PMID 37951571

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the treatment period of Study GA39688/GA39855 and fulfilled the eligibility criteria for the open-label extension (OLE) study were enrolled.
Groups:
- Received Placebo in GA39688 or GA39855; Received Omalizumab in GA39688 or GA39855: After completion of the randomized double-blind placebo controlled studies GA39688 or GA39855, eligible participants were enrolled into WA60169. All participants in WA60169 received 28 weeks of open-label omalizumab as a subcutaneous injection once every 2 weeks (Q2W) or once every 4 weeks (Q4W) before entering a 24-week off-treatment observation phase of the study. Omalizumab dose during the 28 weeks open-label treatment was determined based on serum total IgE levels and body weight from the screening data from the parent studies.
Period: Overall Study
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Started | 126 | 123
Completed | 117 | 114
Not Completed | 9 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 3 | 3
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855 | Total
Number analyzed (Participants) | 126 | 123 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.9) | 49.9 (13.1) | 50.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 82 | 78 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 117 | 110 | 227
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 126 | 117 | 243
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Nasal Polyp Score (NPS)
Description: Total NPS ranges from 0 to 8 (sum of 0-4 for left and right nasal passage scores per the following criteria), with a lower score indicating smaller-sized nasal polyps: 0 = No polyps; 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle turbinate; 2 = Polyps reaching below the lower border of the middle turbinate (modified to accommodate those with a middle turbinectomy, such that polyp must have reached the top of the inferior turbinate.); 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate; and 4 = Large polyps causing complete obstruction of the inferior nasal cavity. Two blinded primary independent expert readers reviewed every post-screening recorded video endoscopy for a given participant to determine total NPS. A third reader chose one of the two scores to be used for analysis in cases where there was any discrepancy in total NPS assigned between the two primary readers.
Time Frame: Baseline, Weeks 4, 8, 16, 24, 36, 52, 64, and 76
Population: Full Analysis Set (FAS) of the open label extension (OLE): all participants enrolled into the OLE, grouped according to the treatment assigned (omalizumab or placebo) at randomization of the previous studies. Participants who were not enrolled in the OLE study, their parent study data were not included in the analyses. All participants in the FAS received at least one dose of study drug.
Measure: Mean (95% Confidence Interval); unit: Sore on a scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Sore on a scale
  Week 4: number analyzed (Participants) | 123 | 121
  Week 4 | -0.17 [-0.38 to 0.05] | -0.85 [-1.07 to -0.63]
  Week 8: number analyzed (Participants) | 126 | 120
  Week 8 | -0.26 [-0.49 to -0.02] | -1.06 [-1.30 to -0.82]
  Week 16: number analyzed (Participants) | 123 | 120
  Week 16 | -0.17 [-0.38 to 0.05] | -1.09 [-1.31 to -0.87]
  Week 24 | -0.19 [-0.42 to 0.03] | -1.01 [-1.24 to -0.78]
  Week 36: number analyzed (Participants) | 120 | 117
  Week 36 | -0.83 [-1.07 to -0.59] | -1.09 [-1.32 to -0.85]
  Week 52: number analyzed (Participants) | 116 | 111
  Week 52 | -0.97 [-1.25 to -0.69] | -1.31 [-1.60 to -1.03]
  Week 64: number analyzed (Participants) | 112 | 110
  Week 64 | -0.40 [-0.66 to -0.13] | -0.85 [-1.12 to -0.58]
  Week 76: number analyzed (Participants) | 109 | 105
  Week 76 | -0.48 [-0.76 to -0.20] | -0.54 [-0.83 to -0.25]

2. Primary Outcome: Change From Baseline in Average Daily Nasal Congestion Score (NCS)
Description: The Nasal Congestion Score (NCS) was assessed daily by the participant via an electronic diary as the response to the following question: Is your nose blocked? The four available response options were scored from 0 (no symptoms) to 3 (severe symptoms): 0 = Not at all; 1 = Mild; 2 = Moderate; and 3 = Severe. For each study day, a score was calculated using an average of the prior 7 days among the available days within the pre-specified window (For Week 24: Study Days 155 to 186), excluding the study day itself, if a value had been recorded by the participant on at least 4 of the prior 7 days; otherwise, the 7-day prior average for that study day was to be considered missing. One calculated (non-missing) 7-day prior average was selected for analysis according to the study day with nearest proximity to Week 24 (Study Day 168), with the earlier selected in the case of a tie. Baseline was defined as the (non-missing) 7-day interval ending on the latest day prior to randomization.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76
Population: FAS-OLE: all participants enrolled into the OLE, grouped according to the treatment assigned (omalizumab or placebo) at randomization of the previous studies. Participants who were not enrolled in the OLE study, their parent study data were not included in the analyses. All participants in the FAS received at least one dose of study drug.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a scale
  Week 4: number analyzed (Participants) | 126 | 122
  Week 4 | -0.17 [-0.27 to -0.07] | -0.39 [-0.50 to -0.29]
  Week 8 | -0.25 [-0.38 to -0.13] | -0.73 [-0.85 to -0.60]
  Week 12 | -0.31 [-0.44 to -0.18] | -0.81 [-0.94 to -0.68]
  Week 16 | -0.32 [-0.46 to -0.19] | -0.88 [-1.02 to -0.74]
  Week 20 | -0.34 [-0.48 to -0.20] | -0.85 [-1.00 to -0.71]
  Week 24 | -0.31 [-0.46 to -0.16] | -0.85 [-1.00 to -0.70]
  Week 28 | -0.61 [-0.76 to -0.47] | -0.88 [-1.03 to -0.73]
  Week 32: number analyzed (Participants) | 124 | 122
  Week 32 | -0.72 [-0.87 to -0.57] | -0.90 [-1.05 to -0.75]
  Week 36: number analyzed (Participants) | 123 | 122
  Week 36 | -0.74 [-0.89 to -0.59] | -0.98 [-1.13 to -0.82]
  Week 40: number analyzed (Participants) | 123 | 120
  Week 40 | -0.73 [-0.88 to -0.59] | -1.02 [-1.17 to -0.87]
  Week 44: number analyzed (Participants) | 123 | 119
  Week 44 | -0.89 [-1.05 to -0.73] | -1.04 [-1.20 to -0.88]
  Week 48: number analyzed (Participants) | 123 | 117
  Week 48 | -0.94 [-1.10 to -0.79] | -1.04 [-1.20 to -0.88]
  Week 52: number analyzed (Participants) | 122 | 116
  Week 52 | -0.99 [-1.14 to -0.83] | -1.12 [-1.28 to -0.96]
  Week 56: number analyzed (Participants) | 121 | 115
  Week 56 | -0.80 [-0.97 to -0.64] | -0.98 [-1.14 to -0.81]
  Week 60: number analyzed (Participants) | 121 | 116
  Week 60 | -0.71 [-0.87 to -0.54] | -0.88 [-1.05 to -0.71]
  Week 64: number analyzed (Participants) | 120 | 117
  Week 64 | -0.63 [-0.80 to -0.46] | -0.88 [-1.05 to -0.71]
  Week 68: number analyzed (Participants) | 118 | 116
  Week 68 | -0.64 [-0.80 to -0.47] | -0.78 [-0.95 to -0.62]
  Week 72: number analyzed (Participants) | 116 | 112
  Week 72 | -0.56 [-0.73 to -0.40] | -0.71 [-0.87 to -0.54]
  Week 76: number analyzed (Participants) | 115 | 111
  Week 76 | -0.58 [-0.76 to -0.41] | -0.65 [-0.83 to -0.48]

3. Primary Outcome: Percentage of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: A serious adverse event was defined as any adverse event that met any of the following criteria: was fatal; was life-threatening; required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the study drug; or, was a significant medical event in the investigator's judgment. Multiple occurrences of the same serious adverse event in one individual were counted once.
Time Frame: From Start to End (Weeks 24 to 52) of OLE Study
Population: All safety analyses were based on the subset of the full analysis set of the OLE study (FAS-OLE), who received at least one dose of omalizumab in the OLE study (Safety-OLE), grouped according to the treatment received (omalizumab or placebo) in the parent studies. One participant randomized to the placebo arm in a parent study accidently received omalizumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 125 | 124
Percentage of Participants
  With at least one AE | 49.6 | 43.5
  With at least one SAE | 4.8 | 2.4

4. Primary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation of Omalizumab
Description: as for outcome 3
Time Frame: From Start to End (Weeks 24 to 76) of OLE Study
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 125 | 124
Percentage of Participants | 0.8 | 0.0

5. Secondary Outcome: Change From Baseline in Average Daily Total Nasal Symptom Score (TNSS)
Description: The Total Nasal Symptom Score (TNSS) was defined as the sum of the four individual scores for Nasal Congestion Score, Anterior Rhinorrhea Score, Posterior Rhinorrhea Score, and Sense of Smell Score, ranging from 0 (no symptoms) to 12 (most severe symptoms), assessed daily by the participant via an electronic diary. For each study day, a score was calculated using an average of the prior 7 days among the available days within the pre-specified window (For Week 24: Study Days 155 to 186), excluding the study day itself, if a value had been recorded by the participant on at least 4 of the prior 7 days; otherwise, the 7-day prior average for that study day was to be considered missing. One calculated (non-missing) 7-day prior average was selected for analysis according to the study day with nearest proximity to Week 24 (Study Day 168), with the earlier selected in the case of a tie. Baseline was defined as the (non-missing) 7-day interval ending on the latest day prior to randomization.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 4: number analyzed (Participants) | 126 | 122
  Week 4 | -0.50 [-0.80 to -0.19] | -1.44 [-1.75 to -1.13]
  Week 8 | -0.72 [-1.09 to -0.34] | -2.44 [-2.82 to -2.06]
  Week 12 | -0.82 [-1.22 to -0.41] | -2.73 [-3.14 to -2.32]
  Week 16 | -0.87 [-1.30 to -0.43] | -2.84 [-3.29 to -2.40]
  Week 20 | -0.93 [-1.36 to -0.49] | -2.84 [-3.27 to -2.40]
  Week 24 | -0.92 [-1.37 to -0.47] | -2.82 [-3.27 to -2.36]
  Week 28 | -1.80 [-2.25 to -1.34] | -2.94 [-3.40 to -2.48]
  Week 32: number analyzed (Participants) | 124 | 122
  Week 32 | -2.19 [-2.64 to -1.74] | -3.14 [-3.60 to -2.68]
  Week 36: number analyzed (Participants) | 123 | 122
  Week 36 | -2.22 [-2.69 to -1.76] | -3.24 [-3.71 to -2.77]
  Week 40: number analyzed (Participants) | 123 | 120
  Week 40 | -2.32 [-2.77 to -1.86] | -3.40 [-3.87 to -2.94]
  Week 44: number analyzed (Participants) | 123 | 119
  Week 44 | -2.72 [-3.21 to -2.24] | -3.52 [-4.02 to -3.03]
  Week 48: number analyzed (Participants) | 123 | 117
  Week 48 | -2.84 [-3.32 to -2.36] | -3.49 [-3.98 to -3.00]
  Week 52: number analyzed (Participants) | 122 | 116
  Week 52 | -3.01 [-3.49 to -2.53] | -3.83 [-4.31 to -3.34]
  Week 56: number analyzed (Participants) | 121 | 115
  Week 56 | -2.54 [-3.04 to -2.04] | -3.23 [-3.74 to -2.72]
  Week 60: number analyzed (Participants) | 121 | 116
  Week 60 | -2.27 [-2.78 to -1.76] | -2.90 [-3.42 to -2.38]
  Week 64: number analyzed (Participants) | 120 | 117
  Week 64 | -1.94 [-2.44 to -1.43] | -2.97 [-3.49 to -2.46]
  Week 68: number analyzed (Participants) | 118 | 116
  Week 68 | -1.83 [-2.33 to -1.33] | -2.59 [-3.09 to -2.08]
  Week 72: number analyzed (Participants) | 116 | 112
  Week 72 | -1.59 [-2.10 to -1.08] | -2.37 [-2.88 to -1.85]
  Week 76: number analyzed (Participants) | 115 | 111
  Week 76 | -1.63 [-2.19 to -1.08] | -2.18 [-2.74 to -1.62]

6. Secondary Outcome: Change From Baseline in Loss of Sense of Smell Score
Description: The Sense of Smell Score was assessed daily by the participant via an electronic diary as the response to the following question: Is your sense of smell reduced? The four available response options were scored from 0 (no symptoms) to 3 (severe symptoms): 0 = Not at all; 1 = Mild; 2 = Moderate; and 3 = Severe. For each study day, a score was calculated using an average of the prior 7 days among the available days within the pre-specified window (For Week 24: Study Days 155 to 186), excluding the study day itself, if a value had been recorded by the participant on at least 4 of the prior 7 days; otherwise, the 7-day prior average for that study day was to be considered missing. One calculated (non-missing) 7-day prior average was selected for analysis according to the study day with nearest proximity to Week 24 (Study Day 168), with the earlier selected in the case of a tie. Baseline was defined as the (non-missing) 7-day interval ending on the latest day prior to randomization.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 4: number analyzed (Participants) | 126 | 122
  Week 4 | -0.07 [-0.16 to 0.02] | -0.22 [-0.31 to -0.13]
  Week 8 | -0.14 [-0.25 to -0.03] | -0.43 [-0.55 to -0.32]
  Week 12 | -0.14 [-0.27 to -0.02] | -0.57 [-0.70 to -0.45]
  Week 16 | -0.19 [-0.33 to -0.06] | -0.58 [-0.72 to -0.44]
  Week 20 | -0.21 [-0.35 to -0.08] | -0.58 [-0.72 to -0.45]
  Week 24 | -0.23 [-0.36 to -0.09] | -0.56 [-0.70 to -0.43]
  Week 28 | -0.26 [-0.40 to -0.12] | -0.58 [-0.72 to -0.44]
  Week 32: number analyzed (Participants) | 124 | 122
  Week 32 | -0.39 [-0.54 to -0.24] | -0.65 [-0.80 to -0.50]
  Week 36: number analyzed (Participants) | 123 | 122
  Week 36 | -0.39 [-0.54 to -0.25] | -0.63 [-0.77 to -0.48]
  Week 40: number analyzed (Participants) | 123 | 120
  Week 40 | -0.42 [-0.57 to -0.27] | -0.66 [-0.81 to -0.51]
  Week 44: number analyzed (Participants) | 123 | 119
  Week 44 | -0.51 [-0.67 to -0.36] | -0.70 [-0.85 to -0.54]
  Week 48: number analyzed (Participants) | 123 | 117
  Week 48 | -0.54 [-0.70 to -0.38] | -0.70 [-0.86 to -0.54]
  Week 52: number analyzed (Participants) | 122 | 116
  Week 52 | -0.60 [-0.76 to -0.43] | -0.76 [-0.92 to -0.59]
  Week 56: number analyzed (Participants) | 121 | 115
  Week 56 | -0.54 [-0.69 to -0.38] | -0.62 [-0.78 to -0.46]
  Week 60: number analyzed (Participants) | 121 | 116
  Week 60 | -0.50 [-0.65 to -0.34] | -0.56 [-0.71 to -0.40]
  Week 64: number analyzed (Participants) | 120 | 117
  Week 64 | -0.41 [-0.57 to -0.26] | -0.53 [-0.68 to -0.37]
  Week 68: number analyzed (Participants) | 118 | 116
  Week 68 | -0.39 [-0.53 to -0.24] | -0.44 [-0.59 to -0.30]
  Week 72: number analyzed (Participants) | 116 | 112
  Week 72 | -0.35 [-0.49 to -0.21] | -0.42 [-0.56 to -0.28]
  Week 76: number analyzed (Participants) | 115 | 111
  Week 76 | -0.35 [-0.50 to -0.20] | -0.39 [-0.54 to -0.24]

7. Secondary Outcome: Change From Baseline in Average Daily Posterior Rhinorrhea Score
Description: The Posterior Rhinorrhea Score was assessed daily by the participant via an electronic diary as the response to the following question: Do you feel dripping at the back of the nose? The four available response options were scored from 0 (no symptoms) to 3 (severe symptoms): 0=Not at all; 1=Mild; 2=Moderate; and 3=Severe. For each study day, a score was calculated using an average of the prior 7 days among available days within a pre-specified window (For Week 24: Study Days 155 to 186), excluding the study day itself, if a value had been recorded by the participant on at least 4 of the prior 7 days, otherwise the 7-day prior average for that study day was to be considered missing. One calculated (non-missing) 7-day prior average was selected for analysis according to the study day with nearest proximity to Week 24 (Study Day 168), with the earlier selected in the case of a tie. Baseline was defined as the (non-missing) 7-day interval ending on the latest day prior to randomization.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 4: number analyzed (Participants) | 126 | 122
  Week 4 | -0.13 [-0.23 to -0.03] | -0.35 [-0.44 to -0.25]
  Week 8 | -0.13 [-0.24 to -0.02] | -0.58 [-0.70 to -0.47]
  Week 12 | -0.14 [-0.25 to -0.02] | -0.60 [-0.72 to -0.48]
  Week 16 | -0.11 [-0.24 to 0.02] | -0.63 [-0.76 to -0.50]
  Week 20 | -0.14 [-0.27 to -0.02] | -0.64 [-0.77 to -0.51]
  Week 24 | -0.15 [-0.29 to -0.02] | -0.66 [-0.79 to -0.52]
  Week 28 | -0.36 [-0.49 to -0.22] | -0.67 [-0.81 to -0.53]
  Week 32: number analyzed (Participants) | 124 | 122
  Week 32 | -0.46 [-0.60 to -0.32] | -0.72 [-0.86 to -0.58]
  Week 36: number analyzed (Participants) | 123 | 122
  Week 36 | -0.46 [-0.60 to -0.32] | -0.76 [-0.90 to -0.62]
  Week 40: number analyzed (Participants) | 123 | 120
  Week 40 | -0.49 [-0.62 to -0.36] | -0.77 [-0.91 to -0.64]
  Week 44: number analyzed (Participants) | 123 | 119
  Week 44 | -0.58 [-0.72 to -0.44] | -0.80 [-0.94 to -0.65]
  Week 48: number analyzed (Participants) | 123 | 117
  Week 48 | -0.60 [-0.74 to -0.46] | -0.77 [-0.91 to -0.62]
  Week 52: number analyzed (Participants) | 122 | 116
  Week 52 | -0.62 [-0.75 to -0.48] | -0.87 [-1.00 to -0.73]
  Week 56: number analyzed (Participants) | 121 | 115
  Week 56 | -0.52 [-0.66 to -0.38] | -0.74 [-0.88 to -0.59]
  Week 60: number analyzed (Participants) | 121 | 116
  Week 60 | -0.47 [-0.62 to -0.33] | -0.70 [-0.85 to -0.55]
  Week 64: number analyzed (Participants) | 120 | 117
  Week 64 | -0.38 [-0.52 to -0.23] | -0.78 [-0.93 to -0.63]
  Week 68: number analyzed (Participants) | 118 | 116
  Week 68 | -0.37 [-0.52 to -0.21] | -0.66 [-0.81 to -0.50]
  Week 72: number analyzed (Participants) | 116 | 112
  Week 72 | -0.27 [-0.42 to -0.11] | -0.61 [-0.76 to -0.45]
  Week 76: number analyzed (Participants) | 115 | 111
  Week 76 | -0.28 [-0.44 to -0.12] | -0.53 [-0.70 to -0.37]

8. Secondary Outcome: Change From Baseline in Average Daily Anterior Rhinorrhea Score
Description: The Anterior Rhinorrhea Score was assessed daily by the participant via an electronic diary as the response to the following question: Do you have a runny nose? The four available response options were scored from 0 (no symptoms) to 3 (severe symptoms): 0=Not at all; 1=Mild; 2=Moderate; and 3=Severe. For each study day, a score was calculated using an average of the prior 7 days among available days within a pre-specified window (For Week 24: Study Days 155 to 186), excluding the study day itself, if a value had been recorded by the participant on at least 4 of the prior 7 days, otherwise the 7-day prior average for that study day was to be considered missing. One calculated (non-missing) 7-day prior average was selected for analysis according to the study day with nearest proximity to Week 24 (Study Day 168), with the earlier selected in the case of a tie. Baseline was defined as the (non-missing) 7-day interval ending on the latest day prior to randomization.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 4: number analyzed (Participants) | 126 | 122
  Week 4 | -0.13 [-0.23 to -0.03] | -0.47 [-0.57 to -0.37]
  Week 8 | -0.21 [-0.32 to -0.09] | -0.68 [-0.80 to -0.57]
  Week 12 | -0.24 [-0.36 to -0.13] | -0.73 [-0.85 to -0.61]
  Week 16 | -0.26 [-0.38 to -0.13] | -0.74 [-0.87 to -0.61]
  Week 20 | -0.24 [-0.37 to -0.11] | -0.74 [-0.87 to -0.61]
  Week 24 | -0.24 [-0.38 to -0.11] | -0.73 [-0.87 to -0.59]
  Week 28 | -0.58 [-0.71 to -0.45] | -0.80 [-0.93 to -0.66]
  Week 32: number analyzed (Participants) | 124 | 122
  Week 32 | -0.65 [-0.77 to -0.52] | -0.84 [-0.97 to -0.71]
  Week 36: number analyzed (Participants) | 123 | 122
  Week 36 | -0.66 [-0.79 to -0.52] | -0.85 [-0.99 to -0.71]
  Week 40: number analyzed (Participants) | 123 | 120
  Week 40 | -0.71 [-0.85 to -0.57] | -0.93 [-1.07 to -0.79]
  Week 44: number analyzed (Participants) | 123 | 119
  Week 44 | -0.77 [-0.91 to -0.63] | -0.96 [-1.10 to -0.82]
  Week 48: number analyzed (Participants) | 123 | 117
  Week 48 | -0.80 [-0.95 to -0.66] | -0.94 [-1.09 to -0.80]
  Week 52: number analyzed (Participants) | 122 | 116
  Week 52 | -0.85 [-0.98 to -0.71] | -1.06 [-1.19 to -0.92]
  Week 56: number analyzed (Participants) | 121 | 115
  Week 56 | -0.71 [-0.85 to -0.56] | -0.89 [-1.03 to -0.74]
  Week 60: number analyzed (Participants) | 121 | 116
  Week 60 | -0.61 [-0.76 to -0.46] | -0.75 [-0.90 to -0.60]
  Week 64: number analyzed (Participants) | 120 | 117
  Week 64 | -0.54 [-0.69 to -0.39] | -0.77 [-0.92 to -0.61]
  Week 68: number analyzed (Participants) | 118 | 116
  Week 68 | -0.47 [-0.62 to -0.32] | -0.69 [-0.84 to -0.54]
  Week 72: number analyzed (Participants) | 116 | 112
  Week 72 | -0.43 [-0.59 to -0.28] | -0.62 [-0.77 to -0.46]
  Week 76: number analyzed (Participants) | 115 | 111
  Week 76 | -0.45 [-0.62 to -0.29] | -0.57 [-0.74 to -0.40]

9. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Assessed by the Total Sino-Nasal Outcome Test (SNOT)-22 Score
Description: The SNOT-22 Questionnaire, a disease specific HRQoL measure, comprises a list of 22 symptoms and social or emotional consequences of the nasal disorder. Every participant was asked to rate how severe each problem had been for them over the past 2 weeks on a scale from 0 (no problem at all) to 5 (problem as bad as it can be). The total score is the sum of the scores for all 22 items, ranging from 0 to 110, with a lower score indicating less disease and better HRQoL. A negative score indicates a decrease (or improvement) from the baseline score.
Time Frame: Baseline, Weeks 4, 8, 16, 24, 36, 52, 64, and 76
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 4: number analyzed (Participants) | 125 | 122
  Week 4 | -8.43 [-10.82 to -6.04] | -17.86 [-20.28 to -15.44]
  Week 8: number analyzed (Participants) | 123 | 122
  Week 8 | -8.85 [-11.56 to -6.15] | -21.74 [-24.47 to -19.01]
  Week 16 | -8.52 [-11.32 to -5.72] | -24.56 [-27.40 to -21.73]
  Week 24: number analyzed (Participants) | 125 | 123
  Week 24 | -7.76 [-10.73 to -4.80] | -23.56 [-26.55 to -20.57]
  Week 36: number analyzed (Participants) | 122 | 118
  Week 36 | -17.87 [-20.91 to -14.83] | -25.42 [-28.51 to -22.34]
  Week 52: number analyzed (Participants) | 119 | 114
  Week 52 | -22.39 [-25.39 to -19.40] | -28.47 [-31.52 to -25.42]
  Week 64: number analyzed (Participants) | 116 | 111
  Week 64 | -17.02 [-20.31 to -13.72] | -22.66 [-26.01 to -19.31]
  Week 76: number analyzed (Participants) | 113 | 112
  Week 76 | -15.37 [-18.79 to -11.95] | -19.44 [-22.89 to -15.99]

10. Secondary Outcome: Change From Baseline in European Quality of Life 5-Dimension 5-Level Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS) Score
Description: The EQ-5D-5L contains a visual analog score (VAS), providing a global assessment of health. The EQ-VAS questionnaire is a self-reported questionnaire that measures health state. The VAS is a 100 mm scale from worst (0 mm) to best (100 mm) health the participant can imagine.
Time Frame: Baseline, Weeks 16, 24, 36, 52, 64, and 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 16: number analyzed (Participants) | 124 | 121
  Week 16 | -0.6 (20.8) | 6.4 (16.7)
  Week 24: number analyzed (Participants) | 125 | 121
  Week 24 | 2.3 (19.6) | 7.9 (16.9)
  Week 36: number analyzed (Participants) | 121 | 117
  Week 36 | 7.4 (20.0) | 9.3 (16.1)
  Week 52: number analyzed (Participants) | 119 | 112
  Week 52 | 8.5 (22.2) | 10.8 (17.9)
  Week 64: number analyzed (Participants) | 116 | 110
  Week 64 | 5.3 (21.4) | 5.3 (18.4)
  Week 76: number analyzed (Participants) | 113 | 110
  Week 76 | 2.8 (20.4) | 4.4 (20.8)

11. Secondary Outcome: Percentage of Participants Reporting "No Problem" in the European Quality of Life 5-Dimension 5-Level Questionnaire (EQ-5D-5L) Subdomains
Description: The EQ-5D-5L contains five domains: Mobility, Self-Care, Usual activity, Pain/Discomfort, and Anxiety/Depression, providing a global assessment of health. Each item is rated by the participant on a five-point scale indicating the followings: Level 1 - no problem; Level 2 - slight problems; Level 3 - moderate problems; Level 4 - severe problems; Level 5 - extreme problems.
Time Frame: Baseline, Weeks 16, 24, 36, 52, 64 and 76
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Percentage of Participants
  Baseline Usual activities: number analyzed (Participants) | 126 | 121
  Baseline Usual activities | 57.9 | 59.5
  Baseline Mobility: number analyzed (Participants) | 126 | 121
  Baseline Mobility | 67.5 | 68.6
  Baseline Self-care: number analyzed (Participants) | 126 | 121
  Baseline Self-care | 83.3 | 90.9
  Baseline Pain/Discomfort: number analyzed (Participants) | 126 | 121
  Baseline Pain/Discomfort | 27.0 | 27.3
  Baseline Anxiety/Depression: number analyzed (Participants) | 126 | 121
  Baseline Anxiety/Depression | 49.2 | 47.9
  Week 16 Usual activities: number analyzed (Participants) | 124 | 123
  Week 16 Usual activities | 54.0 | 75.6
  Week 16 Mobility: number analyzed (Participants) | 124 | 123
  Week 16 Mobility | 60.5 | 79.7
  Week 16 Self-care: number analyzed (Participants) | 124 | 123
  Week 16 Self-care | 84.7 | 91.1
  Week 16 Pain/Discomfort: number analyzed (Participants) | 124 | 123
  Week 16 Pain/Discomfort | 32.3 | 48.0
  Week 16 Anxiety/Depression: number analyzed (Participants) | 124 | 123
  Week 16 Anxiety/Depression | 48.4 | 57.7
  Week 24 Usual activities: number analyzed (Participants) | 125 | 123
  Week 24 Usual activities | 60.8 | 69.9
  Week 24 Mobility: number analyzed (Participants) | 125 | 123
  Week 24 Mobility | 66.4 | 74.0
  Week 24 Self-care: number analyzed (Participants) | 125 | 123
  Week 24 Self-care | 87.2 | 89.4
  Week 24 Pain/Discomfort: number analyzed (Participants) | 125 | 123
  Week 24 Pain/Discomfort | 29.6 | 51.2
  Week 24 Anxiety/Depression: number analyzed (Participants) | 125 | 123
  Week 24 Anxiety/Depression | 47.2 | 60.2
  Week 36 Usual activities: number analyzed (Participants) | 121 | 119
  Week 36 Usual activities | 60.3 | 74.8
  Week 36 Mobility: number analyzed (Participants) | 121 | 119
  Week 36 Mobility | 69.4 | 75.6
  Week 36 Self-care: number analyzed (Participants) | 121 | 119
  Week 36 Self-care | 83.5 | 90.8
  Week 36 Pain/Discomfort: number analyzed (Participants) | 121 | 119
  Week 36 Pain/Discomfort | 40.5 | 48.7
  Week 36 Anxiety/Depression: number analyzed (Participants) | 121 | 119
  Week 36 Anxiety/Depression | 55.4 | 68.9
  Week 52 Usual activities: number analyzed (Participants) | 119 | 114
  Week 52 Usual activities | 65.5 | 74.6
  Week 52 Mobility: number analyzed (Participants) | 119 | 114
  Week 52 Mobility | 72.3 | 71.9
  Week 52 Self-care: number analyzed (Participants) | 119 | 114
  Week 52 Self-care | 87.4 | 91.2
  Week 52 Pain/Discomfort: number analyzed (Participants) | 119 | 114
  Week 52 Pain/Discomfort | 40.3 | 56.1
  Week 52 Anxiety/Depression: number analyzed (Participants) | 119 | 114
  Week 52 Anxiety/Depression | 62.2 | 70.2
  Week 64 Usual activities: number analyzed (Participants) | 116 | 111
  Week 64 Usual activities | 62.9 | 72.1
  Week 64 Mobility: number analyzed (Participants) | 116 | 111
  Week 64 Mobility | 62.1 | 70.3
  Week 64 Self-care: number analyzed (Participants) | 116 | 111
  Week 64 Self-care | 84.5 | 90.1
  Week 64 Pain/Discomfort: number analyzed (Participants) | 116 | 111
  Week 64 Pain/Discomfort | 32.8 | 47.7
  Week 64 Anxiety/Depression: number analyzed (Participants) | 116 | 111
  Week 64 Anxiety/Depression | 50.9 | 61.3
  Week 76 Usual activities: number analyzed (Participants) | 113 | 112
  Week 76 Usual activities | 64.6 | 71.4
  Week 76 Mobility: number analyzed (Participants) | 113 | 112
  Week 76 Mobility | 66.4 | 76.8
  Week 76 Self-care: number analyzed (Participants) | 113 | 112
  Week 76 Self-care | 85.0 | 89.3
  Week 76 Pain/Discomfort: number analyzed (Participants) | 113 | 112
  Week 76 Pain/Discomfort | 34.5 | 48.2
  Week 76 Anxiety/Depression: number analyzed (Participants) | 113 | 112
  Week 76 Anxiety/Depression | 51.3 | 58.0

12. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Score (in Participants With Comorbid Asthma Only)
Description: The AQLQ is a 32-item participant-reported measure of asthma-related quality of life (QoL) with a total score (the mean of all 32 responses) ranging from 1 (severely impaired) to 7 (not impaired at all); a higher score indicates a better QoL. An increase of at least 0.5 points in the AQLQ score was considered the minimal important difference for improvement in QoL.
Time Frame: Baseline, Weeks 16, 24, 36, 52, 64, and 76
Population: FAS-OLE: all participants enrolled into the OLE, grouped according to the treatment assigned (omalizumab or placebo) at randomization of the previous studies. Participants who were not enrolled in the OLE study, their parent study data were not included in the analyses. All participants in the FAS received at least one dose of study drug. Only participants with comorbid asthma were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 69 | 73
Score on a Scale
  Week 16: number analyzed (Participants) | 68 | 69
  Week 16 | 0.05 (1.14) | 0.77 (1.15)
  Week 24: number analyzed (Participants) | 67 | 69
  Week 24 | -0.01 (0.94) | 0.84 (1.25)
  Week 36: number analyzed (Participants) | 67 | 68
  Week 36 | 0.50 (1.05) | 0.84 (1.27)
  Week 52: number analyzed (Participants) | 65 | 62
  Week 52 | 0.52 (1.10) | 0.95 (1.23)
  Week 64: number analyzed (Participants) | 62 | 60
  Week 64 | 0.34 (1.12) | 0.66 (1.35)
  Week 76: number analyzed (Participants) | 61 | 63
  Week 76 | 0.27 (1.15) | 0.42 (1.57)

13. Secondary Outcome: Change From Baseline in Sense of Smell, as Assessed by The University of Pennsylvania Smell Identification Test (UPSIT) Score
Description: The UPSIT is a 40-question instrument that measures an individual's ability to detect odors and ranges from 0 to 40, with a higher score indicating a better sense of smell. It is a self-administered "scratch-and-sniff" test provided in booklets that have 40 microencapsulated odorants, each with a multiple-choice option for the response. The number of correct responses is summed to provide a total score.
Time Frame: Baseline, Weeks 8, 16, 24, 36, 52, 64, and 76
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Score on a Scale
  Week 8: number analyzed (Participants) | 123 | 120
  Week 8 | 0.49 [-0.69 to 1.67] | 5.04 [3.85 to 6.23]
  Week 16: number analyzed (Participants) | 122 | 119
  Week 16 | 0.83 [-0.33 to 1.99] | 4.31 [3.14 to 5.48]
  Week 24: number analyzed (Participants) | 123 | 120
  Week 24 | 0.46 [-0.71 to 1.64] | 4.24 [3.04 to 5.43]
  Week 36: number analyzed (Participants) | 119 | 119
  Week 36 | 3.47 [2.10 to 4.84] | 4.27 [2.90 to 5.65]
  Week 52: number analyzed (Participants) | 116 | 111
  Week 52 | 3.88 [2.57 to 5.20] | 4.13 [2.78 to 5.47]
  Week 64: number analyzed (Participants) | 115 | 109
  Week 64 | 1.81 [0.56 to 3.06] | 2.77 [1.49 to 4.05]
  Week 76: number analyzed (Participants) | 111 | 109
  Week 76 | 0.62 [-0.47 to 1.71] | 1.42 [0.32 to 2.52]

14. Secondary Outcome: Percentage of Participants With a Clinically Significant Change From Baseline in Laboratory Values
Description: Investigators will assess the participants' clinical laboratory values (e.g., serum chemistry, hematology evaluations including complete blood count [CBC] with differential and platelet counts, and urinalysis values) at timepoints throughout this OLE study relative to the participants' values at baseline from studies GA39688/GA39855 and parameters with clinically significant changes from baseline will be reported.
Time Frame: Baseline, Weeks 36, 52, 64, and 76
Population: All safety analyses were based on the subset of the full analysis set of the OLE study (FAS-OLE), who received at least one dose of omalizumab in the OLE study (Safety-OLE), grouped according to the treatment received (omalizumab or placebo) in the parent studies.
Measure: Number; unit: Percentage of Participants
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
Percentage of Participants
  Baseline OLE (Week 24) | 0.0 | 0.0
  Week 36 | 0.0 | 0.0
  Week 52 | 0.0 | 0.0
  Week 64 | 0.0 | 0.0
  Week 76 | 0.0 | 0.0

15. Secondary Outcome: Minimum Serum Concentrations (Ctrough) of Omalizumab at Specified Timepoints
Description: Serum concentrations of omalizumab were quantified using an enzyme-linked immunoabsorbent assay (ELISA) with a lower limit of quantification (LLOQ) of 28.0 nanograms per millilitre (ng/mL). According to the analysis plan, values below the lower limit of quantification (BLQ) were set to 14 ng/mL (i.e. half of LLOQ value). We confirm that all 121 and 123 participants contributed data to the PK outcome measure. The reason why the numbers of participants analyzed per row are different from the overall number of participants is mainly because some PK concentrations at those time points are below LLOQ. Other reasons include: (1) Five participants received accidental dose of Omalizumab at the OLE Week52 thus are excluded for PK sample results for OLE Week64 and OLE Week76, and (2) One participant received omalizumab as concomitant medication in the follow-up period and is excluded from PK sample results for OLE Week76.
Time Frame: Predose at Weeks 36, 52, 64, and 76
Population: The pharmacokinetic evaluable analysis set (PKAS) consisted of participants who received study drug in the form of their per-protocol dose according to baseline total IgE and body weight in the dosing table. Participants receiving the wrong dose or frequency of the treatment assigned (placebo or omalizumab) or the wrong treatment assigned were excluded from this population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 121 | 123
ng/mL
  Week 36: number analyzed (Participants) | 119 | 118
  Week 36 | 33100 (83.8) | 34500 (95.7)
  Week 52: number analyzed (Participants) | 117 | 118
  Week 52 | 29700 (133.4) | 27700 (158.5)
  Week 64: number analyzed (Participants) | 114 | 115
  Week 64 | 1650 (199.8) | 1780 (214.2)
  Week 76: number analyzed (Participants) | 113 | 114
  Week 76 | 93.3 (352.7) | 109 (246.4)

16. Secondary Outcome: Serum Concentration of Total Immunoglobulin E (IgE)
Description: Serum concentrations of total immunoglobulin E (IgE) were measured throughout the study, as target engagement biomarkers of omalizumab, using validated quantitative immunoassays with lower limits of quantification of 2 International Units per millilitre (IU/mL), and upper limits of quantification (ULQ) of 5000 IU/mL.
Time Frame: Predose at Weeks 36, 52, 64, and 76
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
IU/mL
  Week 36 | 665 (530) | 522 (367)
  Week 52 | 635 (463) | 532 (424)
  Week 64 | 390 (366) | 335 (342)
  Week 76 | 231 (226) | 196 (191)

17. Secondary Outcome: Serum Concentration of Free IgE
Description: Serum concentrations of free IgE were measured throughout the study, as target engagement biomarkers of omalizumab, using validated quantitative immunoassays with LLOQ of 0.83 IU/mL, and ULQ of 62.5 IU/mL. The free IgE assay had limited range to measure circulating levels of free IgE in the presence of complexes of omalizumab-IgE. Results above ULQ were set to 62.5 IU/mL. If results for 1/3 or fewer of the participants were greater than the ULQ, then all summary statistics were reported. If the results for more than 1/3 of participants were greater than the ULQ, then only the median, interquartile range and minimum were calculated, and the mean, standard deviation, and maximum were non-reportable.The following are available for median and interquartile ranges (IQR; IQ1-IQ3):
  Placebo: OLE Week 64 median 55.4 (IQR 33.3 - 62.5), OLE Week 76 median 62.5 (IQR 31.1 - 62.5).
  Omalizumab: OLE Week 64 median 55.8 (IQR 37.5 - 62.5), OLE Week 76 median 62.5 (IQR 47.9 - 62.5)
Time Frame: Predose at Weeks 36, 52, 64, and 76
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
Number analyzed (Participants) | 126 | 123
IU/mL
  Week 36: number analyzed (Participants) | 118 | 117
  Week 36 | 8.08 (4.73) | 7.73 (6.37)
  Week 52: number analyzed (Participants) | 117 | 118
  Week 52 | 9.09 (8.81) | 9.52 (10.8)
  Week 64: number analyzed (Participants) | 111 | 112
  Week 64 | NA (NA) — Due to more than 1/3 of the participants having free IgE levels above ULQ, the Mean and SD were not reported (NA) for Weeks 64 and 76. See median and IQR under 'Description', above. | NA (NA) — Due to more than 1/3 of the participants having free IgE levels above ULQ, the Mean and SD were not reported (NA) for Weeks 64 and 76. See median and IQR under 'Description', above.
  Week 76: number analyzed (Participants) | 110 | 113
  Week 76 | NA (NA) — Due to more than 1/3 of the participants having free IgE levels above ULQ, the Mean and SD were not reported (NA) for Weeks 64 and 76. See median and IQR under 'Description', above. | NA (NA) — Due to more than 1/3 of the participants having free IgE levels above ULQ, the Mean and SD were not reported (NA) for Weeks 64 and 76. See median and IQR under 'Description', above.

ADVERSE EVENTS:
Time Frame: From Start to End (Weeks 24 to 76) of OLE Study
Description: All safety analyses were based on the subset of the full analysis set of the OLE study (FAS-OLE), who received at least one dose of omalizumab in the OLE study (Safety-OLE), grouped according to the treatment received (omalizumab or placebo) in the parent studies.
  One participant randomized to the placebo arm in a parent study accidently received omalizumab.
Arm/Group | Received Placebo in GA39688 or GA39855 | Received Omalizumab in GA39688 or GA39855
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/124
Serious Adverse Events (participants affected / at risk) | 12/125 | 8/124
Other Adverse Events (participants affected / at risk) | 28/125 | 19/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Received Placebo in GA39688 or GA39855 (N=125) | Received Omalizumab in GA39688 or GA39855 (N=124)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Testicular abscess (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1/25 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Placebo in GA39688 or GA39855 (N=125) | Received Omalizumab in GA39688 or GA39855 (N=124)
Nasopharyngitis (Infections and infestations) | 13 (34) | 19 (33)
Sinusitis (Infections and infestations) | 13 (16) | 9 (16)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03478930/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03478930/SAP_001.pdf